CLINICAL TRIAL: NCT03019003
Title: A Phase IB Rescue Study With Oral Decitabine (AStX727) and Durvalumab (MEDI4736) Combination Therapy in Recurrent and/or Metastatic Head and Neck Cancer Patients Who Have Progressed on Anti-PD-1, Anti-PD-L1, or Anti-CTLA-4 Monotherapy
Brief Title: Oral Decitabine (ASTX727) and Durvalumab in Recurrent and/or Metastatic Head and Neck Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: AstraZeneca (Industry); Astex Pharmaceuticals, Inc. (Industry)
Responsible Party: Principal Investigator, Sara Pai, MD, PhD, MD, PhD, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-425
Record Dates: First submitted 2017-01-06; First posted 2017-01-12 (Estimated); Results first posted 2025-09-16 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-08

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Decitabine; durvalumab; Azacitidine; tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Oral Decitabine and Durvalumab (Experimental): Oral decitabine (ASTX 727) will be administered alone in Cycle 1 and the combination of oral decitabine and durvalumab therapy will be given in Cycles 2-12.
  Interventions: Drug: Oral Decitabine; Drug: Durvalumab
- 5' Azacitidine 40 mg/m2 on Days 1-5, Durvalumab, and Tremelimumab (Experimental): 5' Azacitidine will be administered alone in Cycle 1 and the combination of 5' Azacitidine, durvalumab, and tremelimumab therapy will be given in Cycles 2-12.
  Interventions: Drug: Durvalumab; Drug: 5' Azacitidine; Drug: Tremelimumab
- 5' Azacitidine 40 mg/m2 on Days 1-5 and 8-12, Durvalumab, and Tremelimumab (Experimental): 5' Azacitidine will be administered alone in Cycle 1 and the combination of 5' Azacitidine, durvalumab, and tremelimumab therapy will be given in Cycles 2-12.
  Interventions: Drug: Durvalumab; Drug: 5' Azacitidine; Drug: Tremelimumab

INTERVENTIONS:
Drug: Oral Decitabine — DNA methyltransferase inhibitor
  Other Names: ASTX 727
  Arms: Oral Decitabine and Durvalumab
Drug: Durvalumab — anti-PD-L1
  Other Names: MEDI4736
Drug: 5' Azacitidine — DNA methyltransferase inhibitor
  Other Names: Vidaza
  Arms: 5' Azacitidine 40 mg/m2 on Days 1-5 and 8-12, Durvalumab, and Tremelimumab; 5' Azacitidine 40 mg/m2 on Days 1-5, Durvalumab, and Tremelimumab
Drug: Tremelimumab — anti-CTLA4
  Arms: 5' Azacitidine 40 mg/m2 on Days 1-5 and 8-12, Durvalumab, and Tremelimumab; 5' Azacitidine 40 mg/m2 on Days 1-5, Durvalumab, and Tremelimumab

SUMMARY:
This is a non-randomized, open-label, Phase Ib study to assess the safety and efficacy of a DNA methyltransferase inhibitor and immune checkpoint inhibitor(s) (durvalumab and/or tremelimumab) combination therapy in the treatment of patients with recurrent and/or metastatic squamous cell carcinoma of the head and neck (SCCHN) who have progressed during or after treatment with anti-PD-1, anti-PD-L1, or anti-CTLA-4 monotherapy for recurrent and/or metastatic disease. The clinical trial is studying drugs that can boost the participant's immune system against the cancer cells as a possible treatment for head and neck cancer.

The study interventions involved in this study are:

* Oral Decitabine (ASTX 727) and 5' Azacytidine
* Durvalumab (MEDI4736) and Tremelimumab

DETAILED DESCRIPTION:
This research study is a Phase I clinical trial, which tests the safety of an investigational drug and also tries to define the appropriate dose of the investigational drug to use for further studies. "Investigational" means that the drugs are still being studied.

The FDA (the U.S. Food and Drug Administration) has not approved durvalumab (MEDI4736) or tremelimumab as a treatment for head and neck cancer.

The FDA (the U.S. Food and Drug Administration) has not approved oral decitabine (ASTX 7272) or 5' Azacytidine for the participant's specific disease but it has been approved for other uses.

This is a first in human study evaluating the safety of combining these different drugs. Durvalumab (MEDI4736) and tremelimumab are part of a family of proteins that make up the immune system. The body generates these proteins, or antibodies, in response to foreign substances (particles not typically found in the body such as bacteria and viruses) and these antibodies can protect against infection. Durvalumab (MEDI4736) and tremelimumab are antibodies that are being studied in several other clinical trials to see if it has an effect in helping the immune system to recognize and eliminate abnormal cells in the body.

Investigators hope that DNA methyltransferase inhibitors may increase the chance of the immune system to recognize the cancer cells.

In this research study, the investigators are looking for the highest effective dose of DNA methyltransferase inhibitors in combination with durvalumab (MEDI4736) and/or tremelimumab to improve the natural ability of the immune system to recognize and target head and neck cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and any locally-required authorization (e.g., HIPAA in the UEU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations
* Age ≥ 18 years at time of study entry or adult male or female (according to age of majority as defined as ≥18 years)
* Histologically confirmed recurrent or metastatic SCCHN (oral cavity, oropharynx, hypopharynx, or larynx) not amenable to therapy with curative intent (surgery or radiation therapy with or without chemotherapy). Patients who refuse radical resection are eligible.
* Tumor progression or recurrence during or after treatment with anti-PD1, anti-PDL1, anti-PDL2, anti-CTLA4, or other immune checkpoint inhibitor where the most recent dose was given within 3 months prior to study registration.
* Must give valid written consent to provide archival FFPE and/or newly acquired tumor tissue for the purpose of establishing baseline PD-L1 status as well as consent to provide on- and/or post-treatment tumor biopsy sample.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 at enrollment
* Life expectancy of > 6 months
* At least 1 lesion that can be accurately measured at baseline as > 10 mm in the longest diameter (except lymph nodes which must have a short axis >15 mm) with CT or MRI and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines.
* Adequate normal organ and marrow function as defined below (within 28 days prior to study registration):

  * Hemoglobin ≥ 9.0 g/dL
  * Absolute neutrophil count (ANC) ≥ 1.5 x 109/L (> 1500 per mm3)
  * Platelet count ≥ 100 x 109/L (>100,000 per mm3)
  * Serum bilirubin ≤ 1.5 x institutional upper limit of normal (ULN). This will not apply to subjects with confirmed Gilbert's syndrome (persistent or recurrent hyperbilirubinemia that is predominantly unconjugated in the absence of hemolysis or hepatic pathology), who will be allowed only in consultation with their physician.
  * AST (SGOT)/ALT (SGPT) ≤ 2.5 x institutional upper limit of normal unless liver metastases are present, in which case it must be ≤ 5x ULN
  * Serum creatinine level <1.5 x ULN and CL>40 mL/min by the Cockcroft-Gault formula (Cockcroft and Gault 1976) or by 24-hour urine collection for determination of creatinine clearance:

Males:

--Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

Females:

--Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)

* Female subjects must either be of non-reproductive potential (ie, post-menopausal by history: ≥60 years old and no menses for ≥1 year without an alternative medical cause; OR history of hysterectomy, OR history of bilateral tubal ligation, OR history of bilateral oophorectomy) or must have a negative serum pregnancy test upon study entry.
* Male subjects with a female partner of childbearing potential must commit to true abstinence from heterosexual contact or commit to the use of male condom plus spermicide throughout the course of the study, and avoid fathering a child during the course of the study (including dose interruptions) and for 6 months following the last dose of azacitidine.
* All men and women of childbearing potential must use acceptable methods of birth control throughout the study as described below:

Females of childbearing potential: Recommendation is for at least one highly effective contraceptive methods during the study and must agree to continue using such precautions for 180 days after the last dose of investigational product.

Non-sterilized males : Non-sterilized male patients who are sexually active with a female partner of childbearing potential must use male condom plus spermicide from screening through 180 days after the last dose of investigational product.

-Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follo

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and/or staff at the study site)
* Histologically confirmed squamous cell carcinoma of any other primary anatomic location in the head and neck (eg. paranasal cavity) and non-squamous histologies (eg. nasopharynx or salivary gland)
* History of another primary malignancy except for:

  * Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of study drug and of low potential risk for recurrence
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease eg, cervical cancer in situ
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 21days prior to the first dose of study drug
* Mean QT interval corrected for heart rate (QTc) ≥470 ms calculated from 3 electrocardiograms (ECGs) using Fredericia's Correction
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab (MEDI4736) or tremelimumab, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid
* Any unresolved toxicity NCI CTCAE grade 2 from previous anti-cancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria.
* Patients with Grade > 2 neuropathy will be evaluated on a case-by-case basis and may be included after consultation with the Study Physician.

  --Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with their assigned IP (eg, hearing loss) may be included after consultation with the Study Physician.
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1
* Abnormal coagulation parameters (PT >15 seconds, PTT>40 seconds, and/or INR >1.5)
* Active or prior documented autoimmune disease within the past 2 years NOTE: Subjects with vitiligo, Grave's disease, or psoriasis not requiring systemic treatment (within the past 2 years) are not excluded.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis)
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to durvalumab (MEDI4736), tremelimumab, or any excipient
* Known or suspected hypersensitivity to azacitidine or mannitol
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, myocardial infarction in the past 6 months, active peptic ulcer disease or gastritis, active bleeding diatheses including any subject known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the subject to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* Uncontrolled systemic fungal, bacterial or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy and/or other treatment)
* History of leptomeningeal carcinomatosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of receiving durvalumab (MEDI4736) or tremelimumab
* Female subjects who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results
* Symptomatic or uncontrolled brain metastases requiring concurrent treatment, inclusive of but not limited to surgery, radiation and/or corticosteroids.
* Subjects with uncontrolled seizures.
* Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 180 days after the last dose of azacitidine, durvalumab (MEDI4736) and/or tremelimumab therapy. Lactating females must agree not to breast feed throughout this period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2024-09-24 (Actual); Study Completion 2024-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Pai, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Qin T, Mattox AK, Campbell JS, Park JC, Shin KY, Li S, Sadow PM, Faquin WC, Micevic G, Daniels AJ, Haddad R, Garris CS, Pittet MJ, Mempel TR, ONeill A, Sartor MA, Pai SI. Epigenetic therapy sensitizes anti-PD-1 refractory head and neck cancers to immunotherapy rechallenge. J Clin Invest. 2025 Mar 17;135(6):e181671. doi: 10.1172/JCI181671. PMID 40091844

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose 5'Aza (40 mg/m^2) for Days 1-5 + Durvalumab + Tremelimumab: Low dose 5'aza (40 mg/m^2) administered subcutaneously daily for 5 days + Durvalumab + Tremelimumab
- Low Dose 5'Aza (40 mg/m^2) for Days 1-5 and 8-12 + Durvalumab 1500 mg Q4W + Tremelimumab 75 mg Q4W: Low dose 5'aza (40 mg/m^2) administered subcutaneously daily for 10 days + Durvalumab + Tremelimumab
- Oral Decitabine 35 mg QD Days 1-3 and Durvalumab 1500 mg Q4W: Oral Decitabine will be administered orally daily for Days 1-3 + Durvalumab 1500 mg Q4W
Period: Overall Study
Arm/Group | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 + Durvalumab + Tremelimumab | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 and 8-12 + Durvalumab 1500 mg Q4W + Tremelimumab 75 mg Q4W | Oral Decitabine 35 mg QD Days 1-3 and Durvalumab 1500 mg Q4W
Started | 7 | 5 | 1
Completed | 7 | 5 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 5' Azacytidine (40 mg/m^2) Days 1-5 + Durvalumab + Tremelimumab; 5' Azacytidine (40 mg/m^2) Days 1-5 and 8-12 + Durvalumab + Tremelimumab: Low Dose 5'aza (40 mg/m^2) SC daily will be administered alone in Cycle 1 and the combination of 5'aza, durvalumab, and tremelimumab therapy will be given in Cycles 2-12.
  5'aza: DNA Methyltransferase Inhibitor
  Durvalumab: anti-PD-L1
  Tremelimumab: anti-CTLA4
- Oral Decitabine Days 1-3 + Durvalumab: Oral Decitabine (35 mg) will be administered alone in Cycle 1 and the combination of decitabine and durvalumab will be given in Cycles 2-12.
  5'aza: DNA Methyltransferase Inhibitor
  Durvalumab: anti-PD-L1
- Total: Total of all reporting groups
Arm/Group | 5' Azacytidine (40 mg/m^2) Days 1-5 + Durvalumab + Tremelimumab | 5' Azacytidine (40 mg/m^2) Days 1-5 and 8-12 + Durvalumab + Tremelimumab | Oral Decitabine Days 1-3 + Durvalumab | Total
Number analyzed (Participants) | 7 | 5 | 1 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 0 | 6
  >=65 years | 4 | 2 | 1 | 7
Age, Continuous [Median (Standard Deviation); unit: years] | 62.9 (6.5) | 61.4 (9.6) | 67.1 (0) | 65.5 (7.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 0 | 1
  Male | 7 | 4 | 1 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 6 | 5 | 1 | 12
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 6 | 4 | 1 | 11
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 7 | 5 | 1 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change in Immune-based Biomarker Expression at Baseline and 2 Months
Description: Greater than 2-fold change in immune-based biomarker expression within the tumor microenvironment
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Groups:
- 5' Azacitidine 40 mg/m^2 on Days 1-5 and 8-12, Durvalumab, and Tremelimumab; 5' Azacitidine 40 mg/m^2 on Days 1-5, Durvalumab, and Tremelimumab: 5' Azacitidine will be administered alone in Cycle 1 and the combination of 5' Azacitidine, durvalumab, and tremelimumab therapy will be given in Cycles 2-12.
  Durvalumab: anti-PD-L1
  5' Azacitidine: DNA methyltransferase inhibitor
  Tremelimumab: anti-CTLA4
Arm/Group | Oral Decitabine and Durvalumab | 5' Azacitidine 40 mg/m^2 on Days 1-5 and 8-12, Durvalumab, and Tremelimumab | 5' Azacitidine 40 mg/m^2 on Days 1-5, Durvalumab, and Tremelimumab
Number analyzed (Participants) | 1 | 5 | 7
Participants | 0 | 1 | 2
Statistical Analysis 1: Comparison: 5' Azacitidine 40 mg/m^2 on Days 1-5 and 8-12, Durvalumab, and Tremelimumab vs 5' Azacitidine 40 mg/m^2 on Days 1-5, Durvalumab, and Tremelimumab; Test type: Other; p < 0.036, t-test, 2 sided

2. Secondary Outcome: Number of Participants With Dose Limiting Toxicity
Description: Adverse events were reported using Common Terminology Criteria for Adverse Events (CTCAE) v4.3.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Decitabine and Durvalumab | 5' Azacitidine 40 mg/m^2 on Days 1-5, Durvalumab, and Tremelimumab | 5' Azacitidine 40 mg/m^2 on Days 1-5 and 8-12, Durvalumab, and Tremelimumab
Number analyzed (Participants) | 1 | 7 | 5
Participants | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored in participants for up to 2 years.
Arm/Group | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 + Durvalumab + Tremelimumab | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 and 8-12 + Durvalumab 1500 mg Q4W + Tremelimumab 75 mg Q4W | Oral Decitabine 35 mg QD Days 1-3 and Durvalumab 1500 mg Q4W
All-Cause Mortality (participants affected / at risk) | 7/7 | 4/5 | 1/1
Serious Adverse Events (participants affected / at risk) | 1/7 | 4/5 | 1/1
Other Adverse Events (participants affected / at risk) | 7/7 | 2/5 | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 + Durvalumab + Tremelimumab (N=7) | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 and 8-12 + Durvalumab 1500 mg Q4W + Tremelimumab 75 mg Q4W (N=5) | Oral Decitabine 35 mg QD Days 1-3 and Durvalumab 1500 mg Q4W (N=1)
Stroke (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Neutropenia (Investigations) | 0 (0) | 1 (1) | 0 (0)
oral hemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 + Durvalumab + Tremelimumab (N=7) | Low Dose 5'Aza (40 mg/m^2) for Days 1-5 and 8-12 + Durvalumab 1500 mg Q4W + Tremelimumab 75 mg Q4W (N=5) | Oral Decitabine 35 mg QD Days 1-3 and Durvalumab 1500 mg Q4W (N=1)
Constipation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
hypomagnesmia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Weight Loss (Investigations) | 2 (2) | 1 (1) | 0 (0)
Pelvic Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Investigations - Other (Investigations) | 4 (4) | 0 (0) | 0 (0)
Alkaline phosphatase increase (Investigations) | 1 (2) | 0 (0) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Aspartate aminotrasnferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
GGT increased (Investigations) | 1 (2) | 0 (0) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Lip Pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 0 (0)
Salivary duct inflammation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Ventricular Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-09-20): https://cdn.clinicaltrials.gov/large-docs/03/NCT03019003/Prot_SAP_000.pdf